CLINICAL TRIAL: NCT00003902
Title: Phase I/II of Capecitabine and Vinorelbine in Elderly Patients (At Least 65 Years) With Metastatic Breast Cancer With or Without Bone Involvement
Brief Title: Capecitabine and Vinorelbine in Treating Older Women Who Have Metastatic Breast Cancer With or Without Bone Involvement
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SAKK 25/99; SWS-SAKK-25/99; EU-99007
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Vinorelbine

INTERVENTIONS:
Drug: capecitabine
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of capecitabine and vinorelbine and to see how well they work in treating older women with metastatic breast cancer with or without bone involvement.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of capecitabine and vinorelbine in elderly women (65 and older) with metastatic breast cancer.
* Evaluate the efficacy and tolerability of this regimen in these patients.
* Assess the time to treatment failure for this regimen as a first line chemotherapy in these patients.

OUTLINE: This is a dose-escalation study of capecitabine and vinorelbine. Patients are stratified according to bone involvement (yes [closed to accrual as of 12/7/04] vs no).

* Phase I: Patients receive oral capecitabine twice daily on days 1-14 and vinorelbine IV over 6-10 minutes on days 1 and 8. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine and vinorelbine until the maximum tolerated dose (MTD) of each drug is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity.

* Phase II: Patients receive capecitabine and vinorelbine administered as in phase I, at the dose preceding the MTD.

Quality of life is assessed during phase II on days 1, 8, and 15 of course 1 and on day 1 of courses 2-4.

Patients are followed every 3 months until disease progression or start of any subsequent antitumor treatment.

PROJECTED ACCRUAL: A total of 98-110 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the breast
* Phase I: Measurable or evaluable disease
* Phase II: Bidimensionally measurable disease
* No CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 65 and over

Sex:

* Female

Menopausal status:

* Postmenopausal

Performance status:

* ECOG/SAKK 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Normal peripheral blood counts

Hepatic:

* AST no greater than 2 times upper limit of normal (ULN) (no greater than 3 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No other prior or concurrent malignancy except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy grade 2 or higher
* No cognitive impairment or severe psychiatric disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* More than 6 months since prior adjuvant chemotherapy
* No prior chemotherapy for metastatic or locally advanced disease
* No other concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapy for metastatic disease allowed
* No continuous concurrent steroids
* No concurrent systemic endocrine therapy for breast cancer
* No other concurrent endocrine therapy

Radiotherapy:

* No concurrent radiotherapy involving greater than 30% of bone marrow or mucosa
* Radiotherapy to nonindicator lesion allowed

Surgery:

* Not specified

Other:

* Bisphosphonates allowed if indicator lesion in nonbone site

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 1999-03; Primary Completion 2004-12 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (phase I)
Response rate at the end of study treatment (phase II)
Toxicity at the end of study treatment (phase II)

SECONDARY OUTCOMES:
Time to treatment failure at end of study treatment (phase II)
Quality of life by Linear Analogue Self-Assessment indicators with 6 assessments until the end of the course 4 (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Hess, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital - St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Hess D, Koberle D, Thurlimann B, Pagani O, Schonenberger A, Mattmann S, Rochlitz C, Rauch D, Schuller JC, Ballabeni P, Ribi K; Swiss Group for Clinical Cancer Research. Capecitabine and vinorelbine as first-line treatment in elderly patients (> or =65 years) with metastatic breast cancer. A phase II trial (SAKK 25/99). Oncology. 2007;73(3-4):228-37. doi: 10.1159/000127414. Epub 2008 Apr 17. PMID 18424887
- [Result] Hess D, Thurlimann B, Pagani O, Aebi S, Rauch D, Ballabeni P, Rufener B, Castiglione-Gertsch M, Goldhirsch A; Swiss Group of Clinical Cancer Research (SAKK). Capecitabine and vinorelbine in elderly patients (> or =65 years) with metastatic breast cancer: a phase I trial (SAKK 25/99). Ann Oncol. 2004 Dec;15(12):1760-5. doi: 10.1093/annonc/mdh467. PMID 15550580